CLINICAL TRIAL: NCT02395003
Title: Study to Investigate Adipocyte Cell and Lipid Turnover in Obese Adolescents
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1503015459; 2R01HD028016-20A1 (NIH); 2R01HD028016 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Pediatric
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — Basal plasma samples for measurements of glucose and glycerol enrichment, and glucose, insulin FFAs, leptin, C-peptide, glucagon, adiponectin, cortisol, growth hormone, catecholamines and amino acids, will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- High VAT/SAT high Palmitate Diet: Subjects with a high ratio of visceral to subcutaneous fat consuming high Palmatite oil diet for 12 weeks
  Interventions: Other: Palmitate Diet
- Low VAT/SAT: Subjects with a low ratio of visceral to subcutaneous fat
  Interventions: Other: Palmitate Diet
- Lean Controls: Lean control
- High VAT/SAT- low Palmitate Diet: Subjects with a high ratio of visceral to subcutaneous fat consuming low Palmatite oil diet for 12 weeks

INTERVENTIONS:
Other: Palmitate Diet — Subject with high VAT/SAT ratio will be randomized to a high or low palmitate oil diet.
  Groups: High VAT/SAT high Palmitate Diet; Low VAT/SAT

SUMMARY:
Insulin Resistance is the best predictor of whether the obese adolescent will develop type 2 diabetes. The present studies will focus on determining what might cause fat to accumulate in the subcutaneous fat regions and lead to local inflammation, causing insulin resistance to develop in obese adolescents.

DETAILED DESCRIPTION:
The purpose of this study is to test whether the reduced transcription of key lipogenic/adipogenic genes in abdominal subcutaneous adipose tissue (SAT) in obese adolescents with a High VAT/SAT (visceral adipose tissue/subcutaneous adipose tissue) ratio translates functionally into a reduced in vivo triglyceride (TG) synthesis and adipocyte proliferation, which in turn will contribute to ectopic fat accumulation and insulin resistance (IR). To test whether the storage capacity of gluteal SAT is linked to the level of VAT/SAT fat distribution in obese adolescents. To explore if changes in dietary fat intake (palmitate intake) alters ceramide concentration in both plasma and adipose tissue (AT) and the Inflammasome complex in the different fat distribution phenotypes and their associations with IR.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (85-95th% age and gender specific) or Obese (>95th% age and gender specific)
* Ages 12-18 years
* Absence of any endocrinopathy
* Absence of any therapy with medication known to alter glucose metabolism (i.e.: Oral steroids, certain psychiatric medications such as Xeleca, Lithium, Paxil)
* English Speaking subjects

Exclusion Criteria:

* Any disease known to alter glucose metabolism (T2DM)
* Diuretic Medication
* Pregnant or breastfeeding
* Type 1 or 2 diabetes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese adolescents
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-04; Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Fat Biopsies | Baseline
  1) To test whether the reduced transcription of key lipogenic/adipogenic genes in abd SAT in obese adolescents with a High VAT/SAT ratio translates functionally into a reduced in vivo TG synthesis and adipocyte proliferation, which in turn will contribute to ectopic fat accumulation and IR.

SECONDARY OUTCOMES:
MRI | Baseline
  Visceral to Subcutaneous fat storage ratio

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No